CLINICAL TRIAL: NCT06315777
Title: Elucidating the GREM1, HAS2 and PTGS2 Gene Expression as Oocytes Development Competency Markers Among Women With Poor Ovarian Reserve (POR) Following the in Vitro Maturation (IVM)
Brief Title: GREM1, HAS2 and PTGS2 Gene Expression Following the in Vitro Maturation (IVM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azrai Abu, Associate Prof, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FRGS/1/2021/SKK01/UKM/02/1
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Increased Oocyte Death; in Vitro Maturation; GREM1 Gene Mutation; Cumulus Cell
Keywords: cumulus cell; GREM 1 gene expression; HAS 2 gene expression; PTGS 2 gene expression; oocyte quality; in vitro maturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal cumulus cell oocytes complex (Experimental): women with normal ovarian reserve will be utilized and analyse the cumulus cell as a baseline
  Interventions: Genetic: cumulus cell oocytes complex (COC) among women with poor ovarian reserve

INTERVENTIONS:
Genetic: cumulus cell oocytes complex (COC) among women with poor ovarian reserve — level of expression of Gremlin-1 (GREM1), Hyaluronic acid synthetase-2 (HAS2), and Prostaglandin-endoperoxide synthase-2 (PTGS2) in cumulus cell oocytes complex (COC) among women with poor ovarian reserve were analyzed

SUMMARY:
Poor ovarian reserve (POR) is an adverse prognostic factor for In-Vitro Fertilization (IVF) success. Numerous established data showed low live birth rates per IVF cycle; 6 to 10%, including the usage of In-Vitro Maturation (IVM). In Malaysia, POR incidence increases mainly from cancer survival, endometriosis, and autoimmune diseases women; therefore, IVM implementation is paramount. In the molecular level, the low competence oocytes showed a low expression of GREM1, HAS2 and PTGS2 in human cumulus cells, thus leading to poor oocyte quality(OQ). Various IVM media had been formulated to enhance the competency and quality of the oocytes to date. Therefore, our study aims to elucidate the GREM1, HAS2 and PTGS2 gene expression as oocyte developmental competency markers among POR women following IVM and tailored to the IVF outcome.

DETAILED DESCRIPTION:
In this study, we will follow up the normal and POR women. The discarded product - cumulus cell will be used in this study for evaluation following the standard IVF cumulus-oocyte-complex denudation. We will develop the In-Vitro Model to assess the expression of GREM1, HAS2, and PTGS2 in normal and POR women first. Subsequently, these gene expressions will be reassessed again via clinical model using IVF-IVM cumulus cell comparing the both groups to elucidate the modifying of oocytes quality following IVM. The cumulus cell RNA will be extracted,and the cDNA will be synthesized and quantitated. The RT-PCR standard curves will be produced, and the concentration range of these genes will be generated and quantified. The OQ, embryo morphology scoring, fertilization rates, and live birth rates will be recorded and compared. We anticipate a higher gene expression associated with good OQ thus better fertilization and live birth rate.

Therefore, this research will understand the impact of IVM in oocytes competency, aiming to improve the fertility rate among POR women in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* women underwent IVF with normal and Poor ovarian reserve based on the Bologna criteria( anti-Müllerian hormone (AMH) below 0.5-1.1 ng/ml]).

Exclusion Criteria:

* Male factor infertility (to reduce bias for embryo quality factor)
* Not agree to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
normal ovarian reserve | for 1 year duration
  the regulation of Gremlin-1 (GREM1), Hyaluronic acid synthetase-2 (HAS2), and Prostaglandin-endoperoxide synthase-2 (PTGS2) in normal cumulus cell oocytes complex (COC).
poor ovarian reserve | for 1 year duration
  the level of expression of Gremlin-1 (GREM1), Hyaluronic acid synthetase-2 (HAS2), and Prostaglandin-endoperoxide synthase-2 (PTGS2) in cumulus cell oocytes complex (COC) among women with poor ovarian reserve

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Reproductive Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Rouhollahi Varnosfaderani S, Hajian M, Jafarpour F, Ghazvini Zadegan F, Nasr-Esfahani MH. Granulosa secreted factors improve the developmental competence of cumulus oocyte complexes from small antral follicles in sheep. PLoS One. 2020 Mar 17;15(3):e0229043. doi: 10.1371/journal.pone.0229043. eCollection 2020. PMID 32182244
- [Result] Anderson RA, Sciorio R, Kinnell H, Bayne RA, Thong KJ, de Sousa PA, Pickering S. Cumulus gene expression as a predictor of human oocyte fertilisation, embryo development and competence to establish a pregnancy. Reproduction. 2009 Oct;138(4):629-37. doi: 10.1530/REP-09-0144. Epub 2009 Jul 14. PMID 19602522
- [Result] McKenzie LJ, Pangas SA, Carson SA, Kovanci E, Cisneros P, Buster JE, Amato P, Matzuk MM. Human cumulus granulosa cell gene expression: a predictor of fertilization and embryo selection in women undergoing IVF. Hum Reprod. 2004 Dec;19(12):2869-74. doi: 10.1093/humrep/deh535. Epub 2004 Oct 7. PMID 15471935
- [Result] Russell DL, Robker RL. Molecular mechanisms of ovulation: co-ordination through the cumulus complex. Hum Reprod Update. 2007 May-Jun;13(3):289-312. doi: 10.1093/humupd/dml062. Epub 2007 Jan 22. PMID 17242016
- [Result] Demiray SB, Goker ENT, Tavmergen E, Yilmaz O, Calimlioglu N, Soykam HO, Oktem G, Sezerman U. Differential gene expression analysis of human cumulus cells. Clin Exp Reprod Med. 2019 Jun;46(2):76-86. doi: 10.5653/cerm.2019.46.2.76. Epub 2019 Jun 1. PMID 31181875
- [Result] Karakaya C, Guzeloglu-Kayisli O, Uyar A, Kallen AN, Babayev E, Bozkurt N, Unsal E, Karabacak O, Seli E. Poor ovarian response in women undergoing in vitro fertilization is associated with altered microRNA expression in cumulus cells. Fertil Steril. 2015 Jun;103(6):1469-76.e1-3. doi: 10.1016/j.fertnstert.2015.02.035. Epub 2015 Apr 22. PMID 25910568